CLINICAL TRIAL: NCT05232292
Title: Influenza Vaccination During COVID19 Outbreak After Acute Coronary Syndrome and Chronic Heart Failure
Brief Title: Influenza Vaccination During Coronavirus Disease 2019 Outbreak After Acute Coronary Syndrome and Chronic Heart Failure
Acronym: IV-ACS&CHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samara Regional Cardiology Dispensary (Other)
Responsible Party: Principal Investigator, Prof. Dmitry Duplyakov FESC, Medical Director, Samara Regional Cardiology Dispensary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOKKD003
Record Dates: First submitted 2021-12-19; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Acute Coronary Syndrome; Chronic Heart Failure
Keywords: acute coronary syndrome; influenza vaccination; prognosis; chronic heart failure
MeSH Terms: conditions — Acute Coronary Syndrome; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccinated (Active Comparator): vaccinated ACS & CHF patients over 65 years
  Interventions: Biological: Ultrix Quadri
- Not vaccinated (No Intervention): not vaccinated ACS & CHF patients over 65 years

INTERVENTIONS:
Biological: Ultrix Quadri — vaccination by Ultrix Quadri against flu
  Arms: Vaccinated

SUMMARY:
Study Description:

Background: Well-known fact that the number of cardiovascular diseases is on the rise during influenza epidemic. It is conceivable that influenza may precipitate plaque rupture, increase cytokines with central roles in plaque destabilization and trigger the coagulation cascade. A number of studies have shown that the risk of cardiovascular complications (ACS, stroke, CHF decompensation, cardiac arrhythmias) seem to be reduced following influenza vaccination. The Influenza Vaccination After Myocardial Infarction study data published in September 2021 have demonstrated a significant decrease of mortality (by 40%) during 1 year of follow-up in patients with myocardial infarction (MI) who has been vaccinated during the first 72 hours.

Objective: the objective is to find out whether influenza vaccination protects against cardiovascular events and death in ACS & CHF patients vaccinated during hospitalization Methods: Population: 400 patients aged 65 and older with acute coronary syndrome are randomized 1:1 and followed up via telephone calls and registries (AIS "Mortality").

Patients will be included in the study in cardiology departments № 1, 2, 3, 5, 6 of the State Budgetary Healthcare Institution "Samara Regional Clinical Cardiology Dispensary named after V.P. Polyakov" Intervention: Influenza vaccination. Control: group of unvaccinated patients. Planned study period is 1 year.

DETAILED DESCRIPTION:
Detailed Description:

Name of investigational treatment: Influenza vaccine ("Ultrix Quadri"™) Planned study period: October - December 2021 ((influenza season) Long-term follow up to 365 days from the moment of vaccination of the last included patient (approximately November-December 2022) via phone calls.

Methodology: vaccination will be start after informed consent on the day of leaving hospital with "Ultrix Quadri"™ vaccine Intervention Model: Parallel Assignment Number of subjects: 400 Number of vaccinated patients is 200 Number of patients with placebo is 200 Primary endpoint: сomposite of all-cause death, MI, or stent thrombosis at 12 months Secondary endpoints

* The number of participants with all-cause death till 1 year (key secondary outcome)
* The number of participants with myocardial infarction till 1 year (key secondary outcome)
* The number of participants with stent thrombosis till 1 year (key secondary outcome)
* The number of participants with cardiovascular death till 1 year (key secondary outcome)
* The number of participants with a new revascularization till 1 year
* The number of participants with cardiovascular death, a new myocardial infarction or stent thrombosis (first occurring) till 1 year
* The number of participants with stroke, including transient ischemic attack (TIA) till 1 year
* The number of participants with hospitalization for heart failure till 1 year
* The number of participants with hospitalization for arrhythmia till 1 year
* Safety of vaccination (incidence of side effects)

Follow up by telephone and registry information (AIS "Mortality"): the follow up for endpoints will be performed using telephone contacts with the patients or first degree relatives.

Purpose of phone calls:

* to assess the safety of vaccination the day after vaccination (T1) 7 (± 1) day after vaccination (T2)
* to study the effectiveness 365 (± 5) days after vaccination (T3)

Reporting for adverse events: The patients will be informed to contact the investigator or study nurse if any adverse event should occur during this timeframe.

Study Start Date: September 2021 Actual Primary Completion Date (safety assessment): December 2021 Actual Study Completion Date (efficiency mark): December 2022 Experimental Drug: influenza vaccine Ultrix Quadri Standard influenza vaccine administered as a deep subcutaneous injection at one occasion per subject.

The experimental drug is not administered to patients in the control group.

Eligibility Criteria:

Ages Eligible for Study: 65 Years and older (Adult, Older Adult) Sexes Eligible for Study: All

Inclusion Criteria:

* Patients with a diagnosis of ACS with transformation to acute MI or unstable angina Patients with a diagnosis of Chronic Heart Failure due to different reasons
* Written informed consent.

Exclusion Criteria:

* Influenza vaccination during the current influenza season or anticipating to be vaccinated during the current influenza season.
* Coronavirus disease 2019 vaccination during 30 days
* Indication for influenza vaccination for some indication other than myocardial infarction.
* Severe allergy to eggs or previous allergic reaction to influence vaccine.
* Suspicion of febrile illness or acute, ongoing infection.
* Hypersensitivity to the active substances or ingredients of Ultrix Quadri or against any residues, such as eggs (ovalbumin or chicken proteins), neomycin, formaldehyde and octoxinol.
* Subjects with endogenic or iatrogenic immunosuppression that may result in reduced immunization response.
* Inability to provide informed consent.
* Age below 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ACS with transformation to AMI or unstable angina
* Patients with a diagnosis of CHF Written informed consent.

Exclusion Criteria:

* • Influenza vaccination during the current influenza season or anticipating to be vaccinated during the current influenza season.

  * COVID-19 vaccination during 30 days
  * Indication for influenza vaccination for some indication other than myocardial infarction.
  * Severe allergy to eggs or previous allergic reaction to influence vaccine.
  * Suspicion of febrile illness or acute, ongoing infection.
  * Hypersensitivity to the active substances or ingredients of Ultrix Quadri or against any residues, such as eggs (ovalbumin or chicken proteins), neomycin, formaldehyde and octoxinol.
  * Subjects with endogenic or iatrogenic immunosuppression that may result in reduced immunization response.
  * Inability to provide informed consent.
  * Age below 65 years.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | up to 1 year
  сomposite of all-cause death, MI, or stent thrombosis at 12 months

SECONDARY OUTCOMES:
Secondary endpoint | up to 1 year
  The number of participants with all-cause death and myocardial infarction till 1 year
Secondary endpoint | 1 week after vaccination
  Safety of vaccination (incidence of side effects)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Duplyakov, Prof, Principal Investigator — SOKKD
Locations (1):
- Samara Regional Cardiology Dispansery, Samara, Russia

IPD SHARING:
Plan to Share IPD: No